CLINICAL TRIAL: NCT03649178
Title: Inflammatory and Vascular Response to Dietary Salt in Rheumatoid Arthritis
Brief Title: Dietary Salt in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, C. Michael Stein, Dan May Professor of Medicine, Professor of Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 141610; R01HL140145 (NIH)
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Salts

STUDY DESIGN:
Intervention Model Description: This will be a random-order, 2 period crossover study with washout
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and nutrition staff will know when participants are on a high salt or low salt diet. Outcomes Assessor will be kept blinded. Participants will be told not to inform outcomes assessor what diet they are on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low salt diet (Other): low-sodium diet (50mmol/24hours x 8 weeks ) Subjects will choose a rotation of low-sodium meals from a predetermined list from a commercial vendor (Mom's Meals) that will be used to provide 2 meals (lunch and dinner)/day that the vendor will deliver at approximately 7 day intervals. Staff of the Vanderbilt Diet,Body Composition, and Human Metabolism Core determine breakfast and snacks appropriate for theHS andLS diets and provide instructions to subjects.
  Interventions: Other: salt
- high salt diet (Other): high-sodium diet (200mmol/24hours x 8weeks) Subjects will choose a rotation of low-sodium meals from a predetermined list from a commercial vendor (Mom's Meals) that will be used to provide 2 meals (lunch and dinner)/day that the vendor will deliver at approximately 7 day intervals. Staff of the Vanderbilt Diet,Body Composition, and Human Metabolism Core determine breakfast and snacks appropriate for theHS andLS diets and provide instructions to subjects.
  Interventions: Other: salt

INTERVENTIONS:
Other: salt — Participants will randomly eat a high salt diet for 8 weeks and a low salt diet for 8 weeks

SUMMARY:
In this study investigators propose to address the following hypotheses: 1) Reduction in dietary sodium will decrease inflammation in patients with rheumatoid arthritis (RA). 2) Reduction in dietary sodium will decrease blood pressure in patients with RA. 3) Reduction in dietary sodium will decrease tissue sodium in patients with RA.

DETAILED DESCRIPTION:
The study is a random-order, 2 period crossover study with washout. Participants will be randomly assigned to be on the high-sodium diet (200mmol/24hours x 8weeks) or low-sodium diet (50mmol/24hours x 8 weeks ) with crossover separated by 4-week washout period. Investigators will allow a 7-day window on the diet (i.e., to facilitate scheduling the diet can be between 7-9 weeks), and investigators will allow a 1-week window for the washout (i.e., washout can be 3-5 weeks).

Investigators will measure changes in inflammation (as measured by DAS28 (using tender and swollen joint count, disease activity and sedimentation rate)), blood pressure measured over a 24 hour period, and tissue sodium (using Magnetic Resonance Imaging (MRI)).

If a relatively simple dietary modification has a clinically important effect on inflammation and blood pressure regulation in vivo in patients with RA, this will have far-reaching implications for the treatment of RA and prevention of Cardiovascular disease in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients older than 18 years who are willing to participate.
2. Satisfy the ACR criteria for the diagnosis of RA.
3. Have stable disease activity as evidenced by no clinically meaningful change in immunomodulating or corticosteroid therapy in the past 1 month.
4. Have moderate disease activity as reflected by a minimum of 3 swollen and tender joints.

Exclusion Criteria:

1. Pregnancy
2. Receiving dialysis
3. Organ or bone marrow transplant
4. Taking diuretics, uncontrolled hypertension (>160/100 mmHg), or cardiac failure requiring treatment.
5. Severe edema (as judged by the investigator)
6. Diabetes mellitus treated with an insulin pump
7. Major surgery within the previous 3 months
8. Severe co-morbid conditions such as active cancer likely to compromise study participation
9. Unwillingness, or other inability, to cooperate
10. Contraindication to MRI
11. Presence of a condition that could make 24-hour blood pressure monitoring difficult: atrial fibrillation, inability to operate machine, receiving anticoagulants, presence of a condition that in the opinion of the investigator may be exacerbated by blood pressure cuff inflation (e.g., lymphedema).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Stein, MBChB, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
all IDP that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: IPD will be shared on request made to the PI. Criteria: Data is not to be shared. Data should only be used for biomedical research. Researchers requesting access will need appropriate IRB approval and sign a data use agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 patients were screened for eligibility between January 2020 to June 2024 at Vanderbilt University Medical Center Rheumatology Clinic.
Pre-assignment Details: 18 of screened participants were randomized. Of the 16 not randomized, 15 did not meet inclusion criteria and 1 declined to participate.
Groups:
- High Sodium Diet, Then Low Sodium Diet: Participants first received high-sodium diet (HSD, 200 mmol/24 hours) for 8 weeks in addition to their baseline DMARD therapy at unchanged doses. After a washout period of 4 weeks, they then received low-sodium diet (LSD, 50 mmol/24 hours) for 8 weeks.
- Low Sodium Diet, Then High Sodium Diet: Participants first received low-sodium diet (LSD, 50 mmol/24 hours) for 8 weeks in addition to their baseline DMARD therapy at unchanged doses. After a washout period of 4 weeks, they then received high-sodium diet (HSD, 200 mmol/24 hours) for 8 weeks.
Period: Overall Study
Arm/Group | High Sodium Diet, Then Low Sodium Diet | Low Sodium Diet, Then High Sodium Diet
Started | 10 | 8
End of First Diet | 9 | 7
Beginning of Second Diet | 8 | 5
Completed | 8 | 4
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — COVID regulation required halt in protocol | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant randomized to sequence A was withdrawn prior to starting diet due to COVID restrictions which halted the study.
Groups:
- Sequence A: High Sodium Diet, Then Low Sodium Diet: A high-sodium diet (200mmol/24hours) will be provided to participants for 8 weeks.
  Then participants will have a 4-week washout in which they eat their typical diet.
  Then a low sodium diet (50mmol/24hours) will be provided to participants for 8 weeks.
- Sequence B: Low Sodium Diet, Then High Sodium Diet: A low sodium diet (50mmol/24hours) will be provided to participants for 8 weeks.
  Then participants will have a 4-week washout in which they eat their typical diet.
  Then a high-sodium diet (200mmol/24hours) will be provided to participants for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Sequence A: High Sodium Diet, Then Low Sodium Diet | Sequence B: Low Sodium Diet, Then High Sodium Diet | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [44 to 62] | 54 [50 to 61] | 55 [50 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17
DAS28-CRP [Median (Inter-Quartile Range); unit: units on a scale] — DAS28-CRP score is a disease activity score based on 28 joints and C-reactive protein. Lower is better. Range= 0.96 units to 10.
  DAS28-CRP = 0.56 x sqrt(tender joint count) + 0.28 x sqrt(swollen joint count) + 0.36 x ln(C-reactive protein + 1) + 0.014 x global health score + 0.96
  units on a scale | 4.8 [4.6 to 5.0] | 5.4 [4.5 to 5.8] | 4.9 [4.5 to 5.5]
Systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 129 [125 to 131] | 118 [114 to 136] | 126 [117 to 133]

OUTCOME MEASURES:

1. Primary Outcome: Change in Tissue Sodium
Description: Investigators will measure change in tissue (skin) sodium using 3.0 T MRI equipped with a 23Na coil.
Time Frame: 2 scans, one at end of week 8, and one at end of week 20
Population: Combined from Sequence A and B.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- High Sodium Diet: This will use data from Sequence A and B after 8 weeks of high sodium (week 8 or 20 depending on sequence).
- Low Sodium Diet: This will use data from Sequence A and B after 8 weeks of low sodium diet (week 8 or 20 depending on sequence).
Arm/Group | High Sodium Diet | Low Sodium Diet
Number analyzed (Participants) | 17 | 17
mmol/L | 17.1 (5.1) | 16.7 (8.2)
Statistical Analysis 1: Comparison: High Sodium Diet; Test type: Other; p = 0.55, Mixed Models Analysis

2. Secondary Outcome: Change in DAS28-CRP
Description: DAS28-CRP score is a disease activity score based on 28 joints and C-reactive protein. Lower is better. Range= 0.96 units to 10.
  DAS28-CRP = 0.56 x sqrt(tender joint count) + 0.28 x sqrt(swollen joint count) + 0.36 x ln(C-reactive protein + 1) + 0.014 x global health score + 0.96
Time Frame: Measured at beginning and end of each diet period at weeks 0, 8, and 12, 20
Population: Combined from Sequence A and B.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- High Sodium Diet Baseline: This will use data from Sequence A and B prior to starting high salt diet (week 0 or 12 depending on sequence).
- High Sodium Diet After 8 Weeks: This will use data from Sequence A and B after 8 weeks of high salt diet (week 8 or 20 depending on sequence).
- Low Sodium Diet Baseline: This will use data from Sequence A and B prior to starting low salt diet (week 0 or 12 depending on sequence).
- Low Sodium Diet After 8 Weeks: This will use data from Sequence A and B after 8 weeks of low salt diet (week 8 or 20 depending on sequence).
Arm/Group | High Sodium Diet Baseline | High Sodium Diet After 8 Weeks | Low Sodium Diet Baseline | Low Sodium Diet After 8 Weeks
Number analyzed (Participants) | 17 | 17 | 17 | 17
units on a scale | 4.50 (0.65) | 4.47 (0.91) | 4.70 (1.21) | 4.21 (1.23)
Statistical Analysis 1: Comparison: High Sodium Diet Baseline; Test type: Other; p = 0.76, Mixed Models Analysis

3. Secondary Outcome: Change in Blood Pressure
Description: Investigators will measure change in systolic blood pressure.
Time Frame: Measured at beginning and end of each diet period at weeks 0,8 and 12, 20
Population: Combined from Sequence A and B.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Sodium Diet Baseline | High Sodium Diet After 8 Weeks | Low Sodium Diet Baseline | Low Sodium Diet After 8 Weeks
Number analyzed (Participants) | 17 | 17 | 17 | 17
mmHg | 125 (10) | 122 (10) | 124 (14) | 114 (11)
Statistical Analysis 1: Comparison: High Sodium Diet Baseline; Test type: Other; p = 0.02, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- High Sodium Diet: This will use data from Sequence A and B during high sodium diet.
- Low Sodium Diet: This will use data from Sequence A and B during low sodium diet.
Arm/Group | High Sodium Diet | Low Sodium Diet
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 3/17 | 7/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Sodium Diet (N=17) | Low Sodium Diet (N=17)
Muscular pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
RA flare (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Baker cyst rupture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Dental infection (Infections and infestations) | 1 (1) | 0 (0)
High blood pressure (Vascular disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was impeded by COVID19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03649178/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT03649178/ICF_000.pdf